CLINICAL TRIAL: NCT02182167
Title: A Randomised Controlled Trial of Intravenous N-acetylcysteine in the Management of Antituberculous Drug-induced Hepatitis
Brief Title: A Trial Of Intravenous N-Acetylcysteine In The Management Of Antituberculous Drug-Induced Hepatitis
Acronym: NAC in TB DIH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Dr Karen Cohen, Dr Karen Cohen, University of Cape Town
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130808; DOH-27-0414-4719. (Registry Identifier: SANCTR)
Record Dates: First submitted 2014-06-18; First posted 2014-07-08 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Drug-Induced Liver Injury
Keywords: Drug Induced Hepatitis (DIH); Toxic Liver; Drug Induced Liver Injury (DILI)
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Acetylcysteine; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV NAC (Experimental): Participants will receive IV N-acetylcysteine or placebo. The dosing regimen is based on the regimens used in paracetamol poisoning .
  Initial dose: 150 mg/kg body mass of N-acetylcysteine/WFI infused in 200 mL of 5% dextrose intravenously over 60 minutes, followed by continuous infusion: 50 mg/kg body mass in 500 mL of 5% dextrose over next 4 hours, followed by 100 mg/kg body mass in 1 litre of 5% dextrose over 16 hours.
  Interventions: Drug: IV N-acetylcysteine (NAC)
- Placebo (Placebo Comparator): Water
  Interventions: Drug: Water

INTERVENTIONS:
Drug: IV N-acetylcysteine (NAC)
  Other Names: Paradote
  Arms: IV NAC
Drug: Water
  Arms: Placebo

SUMMARY:
We will conduct a randomized placebo controlled trial to determine whether administration of intravenous (IV) NAC to participants with TB DIH, in dosages similar to that used in paracetamol poisoning, can improve recovery from hepatotoxicity.

DETAILED DESCRIPTION:
South Africa has a huge tuberculosis (TB) disease burden, with 948 per 100 000 people diagnosed with TB in 2008. TB drug induced hepatitis (DIH) is a common adverse effect of TB therapy that causes significant patient morbidity and prolonged hospital stays. N-Acetylcysteine (NAC) has been extensively studied and used for many years in the treatment of paracetamol-induced hepatotoxicity, with good evidence of efficacy and safety. NAC has also been used in other forms of liver injury and drug toxicity. It has not previously been used in the management of TB DIH.

We will screen all patients with clinical hepatitis on TB treatment admitted to New Somerset and Groote Schuur hospitals and aim to recruit 100 participants over 3 years. We will randomise 50 participants to receive an IV loading dose of 150mg/kg of NAC over 60 minutes followed by 50mg/kg IV over 4 hours by continuous infusion and finally 100mg/kg IV over 16 hours. Fifty participants will be randomised to receive placebo. The primary outcome will be time to normalisation of liver function (ALT<100). We will also determine the effect of NAC on duration of hospitalization, rate of recovery from liver failure, all cause mortality, and describe adverse effects of IV NAC in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old
* Diagnosed with pulmonary or extrapulmonary tuberculosis based on symptoms, radiological features and/or laboratory evidence.
* On first line antituberculous therapy
* Diagnosed with TB DIH

Exclusion Criteria:

* Patients with a diagnosis of acute viral hepatitis based on a positive anti-HAV, IgM, anti- HBcIgM, or confirmed hepatitis C infection
* Patients known to be asthmatic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
ALT normalisation | up to 8 weeks
  To determine the effect of IV NAC on the time to normalization of liver function in patients with TB DIH

SECONDARY OUTCOMES:
Duration of hospitalization | up to 8 weeks
  To determine the effect of IV NAC on duration of hospitalization
Recovery from liver failure | up to 8 weeks
  To determine the effect of IV NAC on the rate of recovery from liver failure
All-cause mortality | up to 8 weeks
  To determine the effect of IV NAC on all-cause mortality in patients with TB DIH
Adverse Events | up to 8 weeks
  To determine the adverse event profile of IV NAC when administered to patients with TB DIH
TB Drug Rechallenge | up to 8 weeks
  To determine the effect of IV NAC on success of TB drug rechallenge.
Rechallenge duration | up to 8 weeks
  To determine the effect of IV NAC on duration of rechallenge

OTHER OUTCOMES:
Biomarkers
  To store blood, urine and biopsy specimens (if biopsies were taken as part of patient management),bank serum, to enable us to conduct future sub studies exploring mechanisms, predictors and biomarkers of TB DIH, genetic associations with TB DIH and improved diagnostic strategies

CONTACTS AND LOCATIONS:
Overall Officials: Karen Cohen, Principal Investigator — University of Cape Town
Locations (2):
- South Africa (2):
  - Groote Schuur Hospital, Cape Town, Western Province
  - New Somerset Hospital, Cape Town, Western Province